CLINICAL TRIAL: NCT02285075
Title: A Clinical Pharmacokinetic Study: Is Three Times Weekly Temocillin Appropriate for the Treatment of Severe Gram-negative Infections in Patients With ESRD Treated With Intermittent Hemodialysis?
Brief Title: Temocillin Pharmacokinetic in Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Collaborators: Paul Tulkens, Louvain drug research institute, belgium (Unknown); Francoise Van Bambeke, Louvain drug research institute, belgium (Unknown); Ana Miranda Bastos, Louvain drug research institute, belgium (Unknown)
Responsible Party: Principal Investigator, Vandecasteele Stefaan Johan, Stefaan Johan Vandecasteele, MD, PhD, AZ Sint-Jan AV
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVDC Temocillin 1
Record Dates: First submitted 2014-11-02; First posted 2014-11-06 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Gram-Negative Bacterial Infections; Renal Failure Chronic Requiring Hemodialysis
Keywords: temocillin; PD/PD; T>MIC
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- temocillin PK/PD in haemodialysis (Other): Pharmacokinetic study measuring total and free temocillin concentrations in patients treated with haemodialysis receiving 1 gram temocillin for a 1 day interval, 2 gram temocillin for a two day interval and 3 gram temocillin for a 3 day interval to the next dialysis session
  Interventions: Drug: temocillin PK/PD in haemodialysis

INTERVENTIONS:
Drug: temocillin PK/PD in haemodialysis — Pharmacokinetic study measuring total and free temocillin concentrations just before, and at 0.5, 3, 6, 12, 20 (before dialysis) and 24 (at the end of dialysis) hours after start of the infusion when patients were dialysed with a 1-day interval; just before and at 0.5, 3, 6, 12, 24, 36, 44 (before dialysis) and 48 (at the end of dialysis) hours after start of the infusion when patients were dialysed with a 2-day interval, and just before and at 0.5, 3, 6, 12, 24, 36, 48, 68 (before dialysis) and 72 (at the end of dialysis) hours after start of the infusion if patients were dialysed with a 3-day interval in order to determine basic PK and PD parameters in patients treated with intermittent haemodialysis and temocillin (Vd, T1/2, protein binding, clearance, reduction rate and T > MIC of 8 and 16 mg/L).

SUMMARY:
The current study aimed to explore the pharmacokinetics of temocillin in patients treated with haemodialysis and to demonstrated whether or not the pharmacodynamics target of a time above a MIC of 16 mg/L of more than 40 and 60 % of the dosing interval could be obtained with a dosing schedule of 1 gram/24 hours, 2 gram/48 hours and 3 gram/72 hours, all of these doses given after haemodialysis sessions only.

DETAILED DESCRIPTION:
Background: Temocillin is a renally cleared penicillin with long serum half-live and potent activity against most gram-negative bacteria, making it an ideal candidate for treatment given on dialysis days only of severe gram-negative infections in patients with ESRD treated with haemodialysis.

Endpoints:

Primary: The current study aimed to demonstrated by measurement of AUC whether or not the pharmacodynamics target of a time above a MIC of 8 and 16 mg/L of more than 40 and 60 % of the dosing interval could be obtained with a dosing schedule of 1 gram/24 hours, 2 gram/48 hours and 3 gram/72 hours, all of these doses given after haemodialysis sessions only.

Secondary: Key pharmacokinetic and dialytic parameters were determined as previously described16. The following parameters were recorded: the volume of distribution Vd (determined as Vd = dose / (Tempeak - Temtrough) in liter); the Vd/Wt (in liter/kg body weight); the non-dialysis clearance of temocillin (Ke(non-dialysis) = [ln(Tempeak) - ln(Tempre)] / time between peak level and start of next dialysis); the non-dialysis half-life (T1/2(non-dialysis) = 0.693 / Ke(non-dialysis) in hours); the dialysis clearance of temocillin (Ke(dialysis) = [ln(Tempre) - ln(Tempost)] / dialysis duration); the dialysis half-life (T1/2(dialysis) = 0.693 / Ke(dialysis) in hours); the Urea Reduction Ratio (URR = (BUNpre - BUNpost) / BUNpre); the Temocillin Reduction Ratio TRR = (Tempre - Tempost) / Tempre); the Temocillin Removal Ratio (the total amount of temocillin recovered in the dialysate, based on the area under the curve of the temocillin removal rate and the treatment time); and the AUC of temocillin. For all PK/PD analysis, the non-compartmental method using RStudio 0.98.501 with R 3.0.2 software was used.

Methods: Pharmacokinetic study measuring total and free temocillin concentrations in patients treated with intermittent haemodialysis and temocillin. Blood samples were drawn just before, and at 0.5, 3, 6, 12, 20 (before dialysis) and 24 (at the end of dialysis) hours after start of the infusion when patients were dialysed with a 1-day interval; just before and at 0.5, 3, 6, 12, 24, 36, 44 (before dialysis) and 48 (at the end of dialysis) hours after start of the infusion when patients were dialysed with a 2-day interval, and just before and at 0.5, 3, 6, 12, 24, 36, 48, 68 (before dialysis) and 72 (at the end of dialysis) hours after start of the infusion if patients were dialysed with a 3-day interval. Patients were followed for 1 to 6 subsequent AUC. Dialysate samples were taken 1, 2, 3 and 4 h after the start of dialysis. All samples were taken from an arterial or venous catheter, after thorough rinsing. Serum (obtained by centrifugation after blood clotting) and dialysate was frozen (-80 C) immediately after sampling until analysis.

Temocillin total and free concentrations were determined with high performance liquid chromotography(HPLC) with a LiChrospher 100 RP-18 5 μm column (Merck AG), using an elution buffer 100 mM Na acetate buffer pH 7/acetonitrile (95:5, v/v), a flow rate 1 mL/min and a Waters 2690 Alliance System (Waters Corp., Milford, MA, USA), with quantification at 235 nm as previously described.

ELIGIBILITY:
Inclusion Criteria:

* all patients under treatment with haemodialysis for ESRD for whom a treatment with temocillin was indicated according to the attending physician were eligible for the study.

Exclusion Criteria:

* an age of less than 18 years
* an estimated life-expectance of < 24 hours due to major co-morbid conditions
* pregnancy
* an IgE-mediated allergy to penicillins
* patients not giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
% of the dosing interval time above an MIC of 8 and 16 mg/L (% T>MIC 8 or 16 mg/L) | two to ten days
  Is T > MIC 8 and 16 mg/ML > 40 or 60 %

SECONDARY OUTCOMES:
Determine basic pharmacokinetic parameters of temocillin in intermittent haemodialysis | two to ten days
  Vd (volume of distribution)
Determine basic pharmacokinetic parameters of temocillin in intermittent haemodialysis | two to ten days
  T1/2 (serum half life, on and of dialysis)
Determine basic pharmacokinetic parameters of temocillin in intermittent haemodialysis | two to ten days
  Temocillin clearance (renal and non-renal)
Determine basic pharmacokinetic parameters of temocillin in intermittent haemodialysis | two to ten days
  Temocillin reduction rate
Determine basic pharmacokinetic parameters of temocillin in intermittent haemodialysis | two to ten days
  temocillin removal rate
Determine basic pharmacokinetic parameters of temocillin in intermittent haemodialysis | two to ten days
  temocillin protein binding

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan J Vandecasteele, MD, PhD, Principal Investigator — AZ Sint-Jan AV
Locations (2):
- Belgium (2):
  - AZ Sint-Jan Brugge Oostende AV, Bruges
  - Louvain Drug Research Institute (LDRI), Brussels

REFERENCES:
- [Result] Miranda Bastos AC, Vandecasteele SJ, Tulkens PM, Spinewine A, Van Bambeke F. Development and validation of a high performance liquid chromatography assay for the determination of temocillin in serum of haemodialysis patients. J Pharm Biomed Anal. 2014 Mar;90:192-7. doi: 10.1016/j.jpba.2013.12.002. Epub 2013 Dec 12. PMID 24389461
- [Derived] Miranda Bastos AC, Vandecasteele SJ, Spinewine A, Tulkens PM, Van Bambeke F. Temocillin dosing in haemodialysis patients based on population pharmacokinetics of total and unbound concentrations and Monte Carlo simulations. J Antimicrob Chemother. 2018 Jun 1;73(6):1630-1638. doi: 10.1093/jac/dky078. PMID 29579214